CLINICAL TRIAL: NCT06423443
Title: Digital Cognitive Behavioral Therapy for Depressive Disorders: A Randomized Controlled Trial
Brief Title: Digital Cognitive Behavioral Therapy for Depressive Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Adai Technology (Beijing) Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ICBT2301
Record Dates: First submitted 2024-05-16; First posted 2024-05-21 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Cognitive Behavioral Therapy (Experimental)
  Interventions: Behavioral: Digital Cognitive Behavioral Therapy; Drug: TAU
- Health Education (Active Comparator)
  Interventions: Behavioral: Health Education; Drug: TAU

INTERVENTIONS:
Behavioral: Digital Cognitive Behavioral Therapy — digital cognitive behavioral therapy app
  Arms: Digital Cognitive Behavioral Therapy
Behavioral: Health Education — traditional on-line health education app
  Arms: Health Education
Drug: TAU — treatment as usual

SUMMARY:
This study aims to explore the effectiveness of digital interventions combined with medication in the treatment of patients with depressive disorders. Its main aim is to answer: Can digital interventions combined with medication effectively alleviate symptoms of depression? The experiment will compare the effects of medication combined with digital interventions to those combined with online mental health education to evaluate their relative effectiveness. Participants will be required to engage with the medication plus digital therapy for a duration of two months, and follow-up assessments will be conducted to evaluate the long-term effects of the treatments and monitor any changes in depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Meets the diagnostic criteria for depression according to the DSM-5 (Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition), without psychotic symptoms, as recurrent outpatient or inpatient.
2. Patients with a Montgomery-Asberg Depression Rating Scale (MADRS) score ≥ 22 before randomization.
3. Age ≥ 18 and ≤ 65 years, regardless of gender.
4. Understands the trial and signs the informed consent form.

Exclusion Criteria:

1. Meets criteria for other psychiatric disorders according to the DSM-5, including schizophrenia spectrum disorders, bipolar and related disorders, neurodevelopmental disorders, neurocognitive disorders, or depression due to substance and/or medication or other medical conditions.
2. History of substance and/or alcohol abuse within the past year.
3. Significant risk of suicide (MADRS item 10 score = 4).
4. Difficulty or inability to communicate verbally, understand or follow instructions, or cooperate with treatment and assessment.
5. Inability to use a smartphone.
6. Deemed unsuitable for participation by the researcher.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS) | baseline and immediately after 8-week intervention, and follow-ups at 4 weeks, 12 weeks, and 6 months
  Score Range: 0 (best outcome) to 60 (worst outcome) Higher scores indicate worse depression symptoms.

SECONDARY OUTCOMES:
PHQ-9 (Patient Health Questionnaire-9) | baseline and weekly assessments during the treatment period, assessed up to 8 weeks, and follow-ups at 4 weeks, 12 weeks, and 6 months
  PHQ-9 Score Range: 0 (best outcome) to 27 (worst outcome); higher scores indicate more severe depression symptoms.
GAD-7 (Generalized Anxiety Disorder-7) | baseline and weekly assessments during the treatment period, assessed up to 8 weeks, and follow-ups at 4 weeks, 12 weeks, and 6 months
  GAD-7 Score Range: 0 (best outcome) to 21 (worst outcome); higher scores indicate more severe generalized anxiety symptoms.
Snaith-Hamilton Pleasure Scale (SHAPS) | baseline, immediately after 8-week intervention, and follow-ups at 4 weeks, 12 weeks, and 6 months
  Score Range: 14 (best outcome) to 56 (worst outcome) Higher scores indicate greater levels of anhedonia (reduced ability to experience pleasure).
Rumination Response Scale (RRS) | baseline, immediately after 8-week intervention, and follow-ups at 4 weeks, 12 weeks, and 6 months
  Score Range: 22 (best outcome) to 88 (worst outcome) Higher scores indicate higher levels of rumination.
Pittsburgh Sleep Quality Index (PSQI) | baseline, immediately after 8-week intervention, and follow-ups at 4 weeks, 12 weeks, and 6 months
  Score Range: 0 (best outcome) to 21 (worst outcome) Higher scores indicate poorer sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Chengdu, Sichuang, China